CLINICAL TRIAL: NCT00180128
Title: AIDA2000 - Risk-Adapted Therapy for Patients With Acute Promyelocytic Leukemia(APL)
Brief Title: AIDA2000 - Risk-Adapted Therapy for Patients With Acute Promyelocytic Leukemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Prof. Dr. Gerhard Ehninger, Dresden University of Technology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MK1-192
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-07

CONDITIONS: Leukemia, Promyelocytic, Acute
Keywords: acute promyelocytic leukemia; risk adapted therapy
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Idarubicin; Mitoxantrone; Daunorubicin; Cytarabine

INTERVENTIONS:
Drug: all-trans retinoid acid
Drug: idarubicin
Drug: mitoxantrone
Drug: daunorubicin
Drug: cytarabine

SUMMARY:
In AIDA 2000 therapy of acute promyelocytic leukemia (APL) is given in a risk-adapted manner. Risk factors are age and white-blood-cell (WBC)-count at diagnosis. Induction therapy is done with ATRA and idarubicin followed by postremission therapy with daunorubicin and mitoxantrone in age adapted dosages. Patients with an high WBC were additionally treated with cytarabine. Finally a two year period of maintenance therapy with 6-mercaptopurine, methotrexate and ATRA is performed.

DETAILED DESCRIPTION:
In AIDA 2000 therapy of acute promyelocytic leukemia (APL) is given in a risk-adapted manner. Risk factors are age and white-blood-cell (WBC)-count at diagnosis. Induction therapy is done with ATRA and idarubicin followed by postremission therapy with daunorubicin and mitoxantrone in age adapted dosages. Patients with an high WBC were additionally treated with cytarabine. Finally a two year period of maintenance therapy with 6-mercaptopurine, methotrexate and ATRA is performed.

ELIGIBILITY:
Inclusion Criteria:

* acute promyelocytic leukemia confirmed by detection of t(15;17) and/or PML/RARa
* no contraindication for chemotherapy
* written informed consent

Exclusion Criteria:

- severe comorbidities

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2000-01; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
overall survival

SECONDARY OUTCOMES:
toxicity of the regimen
evaluation of additional risk factors
effectiveness of MRD as guidance for therapy decisions
relapse free survival
complete remission rate

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Ehninger, MD, Principal Investigator — Department of Medicine I, University Hospital Carl Gustav Carus Dresden
Locations (1):
- Department of Medicine I, University Hospital Carl Gustav Carus, Dresden, Germany